CLINICAL TRIAL: NCT01494181
Title: Postoperative Vascular Events in Unrecognised Obstructive Sleep Apnea
Brief Title: Unrecognised Obstructive Sleep Apnea Study
Acronym: OSA
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Other Study IDs: Version Nov 14, 2011
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; vascular events
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Plan of investigation:

This is an observational cohort study to determine the effect of OSA, independent of other risk factors, on postoperative vascular events. The study is conceived, designed and will be conducted, and analyzed independent to any company. There is no commercial sponsorship.

DETAILED DESCRIPTION:
The potential study subjects will be approached by study coordinator at preoperative clinic. If the patient is interested in participating the study, he/she will be screened and consented. Undetected or untreated OSA will be established by STOP-Bang questionnaire and subsequent overnight PSG by using Apnea Link Plus which is level ( 2 ) at patient's home.The following data will be recorded: including age, gender, history of coronary artery disease, prior revascularization, cerebrovascular disease, peripheral vascular disease, critical aortic valvular stenosis, congestive heart failure, atrial fibrillation, diabetes treated with insulin or an oral diabetic drug, hypertension, hypercholesterolemia treated with drug therapy, tobacco use, renal insufficiency and the type of surgery. For all study patients, the nocturnal blood oxygen saturation will be monitored by a pulse oximeter (PULSOX 300i) for first 3 nights postoperatively.During their stay in hospital, patients will be followed daily, and outcomes will be recorded, until discharge.. ECG will be measured preoperatively and repeated on day 1 to 3 after surgery. Venous blood will be collected 6-12 hours and on the first 3 days after surgery for measuring cTnT concentration.If patient's ECG is abnormal and/or patient is positive for troponin test, treating physician will be contacted for further treatment. Patient will be contacted 30 days after surgery by phone to ascertain if they have experienced any adverse out come.

ELIGIBILITY:
Patients Inclusion & Exclusion Criteria:

Inclusion criteria:

Ethics Committee approval and informed consent will be obtained. We plan to study patients at moderate-to-high risk for postoperative vascular complications because our data from other trials suggested that the incidence of OSA in these patients is higher than the general population. We will include patients who are:

1. adult males and females, age ≥ 45 years, undergoing elective non-cardiac surgery that is expected to require a postoperative hospital stay of more than 3 nights, and
2. at increased risk for postoperative vascular events, defined as having at least one of the following risk factors (a) high-risk surgery (intra-peritoneal, intra-thoracic or supra-inguinal vascular surgery); (b) history of ischemic heart disease; (c) history of congestive heart failure; (d) history of cerebrovascular disease (d) diabetes requiring insulin therapy (e) serum creatinine > 175 µmol/L.

Exclusion criteria:

Patients will be excluded if:

1. they have a previous diagnosis of OSA or any sleep-related breathing disorder and on treatment
2. they are unwilling or physically unavailable for PSG on any night before surgery;
3. their surgery included tonsillectomy, septoplasty, uvuloplasty, pharyngoplasty, tracheostomy, or prolonged (> 48 hrs) postoperative mechanical ventilation of the lungs is anticipated. It is because these procedures/interventions are likely to cure or at least modify the severity of OSA.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patient
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2011-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
primary outcome of this study is postoperative vascular event within 30 days after surgery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (4):
- The Scarborough hospital, Scarborough Village, Ontario, Canada
- Prince of Wales Hospital, Shatin, Hong Kong
- Unversity Malaya Medical Centre, Kuala Lumpur, Malaysia
- Khoo Teck Puat Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Chung F, Waseem R, Wang CY, Seet E, Suen C, Chan MTV; Postoperative Vascular Complications in Unrecognised Obstructive Sleep Apnea (POSA) Study Investigators. Preoperative oximetry-derived hypoxemia predicts postoperative cardiovascular events in surgical patients with unrecognized obstructive sleep apnea. J Clin Anesth. 2022 Jun;78:110653. doi: 10.1016/j.jclinane.2022.110653. Epub 2022 Feb 4. PMID 35131555
- [Derived] Seet E, Chung F, Wang CY, Tam S, Kumar CM, Ubeynarayana CU, Yim CC, Chew EFF, Lam CKM, Cheng BCP, Chan MTV. Association of Obstructive Sleep Apnea With Difficult Intubation: Prospective Multicenter Observational Cohort Study. Anesth Analg. 2021 Jul 1;133(1):196-204. doi: 10.1213/ANE.0000000000005479. PMID 33720906
- [Derived] Waseem R, Chan MTV, Wang CY, Seet E, Tam S, Loo SY, Lam CKM, Hui DS, Chung F. Diagnostic performance of the STOP-Bang questionnaire as a screening tool for obstructive sleep apnea in different ethnic groups. J Clin Sleep Med. 2021 Mar 1;17(3):521-532. doi: 10.5664/jcsm.8940. PMID 33112227
- [Derived] Chan MT, Wang CY, Seet E, Tam S, Lai HY, Walker S, Short TG, Halliwell R, Chung F; POSA Investigators. Postoperative vascular complications in unrecognised Obstructive Sleep apnoea (POSA) study protocol: an observational cohort study in moderate-to-high risk patients undergoing non-cardiac surgery. BMJ Open. 2014 Jan 9;4(1):e004097. doi: 10.1136/bmjopen-2013-004097. PMID 24413351